CLINICAL TRIAL: NCT02729740
Title: SMART - A Prospective, Multicenter Registry Assessing the Embolization of Neurovascular Lesions Using the Penumbra SMART COIL® System
Brief Title: Assessment of the Embolization of Neurovascular Lesions Using the Penumbra Smart Coil
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 10023
Record Dates: First submitted 2016-03-15; First posted 2016-04-06 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Intracranial Aneurysm
Keywords: Penumbra Smart coils; PC 400; AV malformations; AV fistulae; POD
MeSH Terms: conditions — Intracranial Aneurysm; Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Penumbra Smart System (Other)
  Interventions: Device: Penumbra Smart Coil; Device: Penumbra Coil 400TM (PC400), Penumbra Occlusion DeviceTM(POD)

INTERVENTIONS:
Device: Penumbra Smart Coil
Device: Penumbra Coil 400TM (PC400), Penumbra Occlusion DeviceTM(POD) — Other Penumbra Coils available as standard of care

SUMMARY:
The primary objective of this study is to gather post market data on the Penumbra SMART COIL® System (Smart System) in the treatment of intracranial aneurysms and other malformations.

DETAILED DESCRIPTION:
This is a prospective, multi-center registry of patients treated in accordance with the cleared indications for the Smart System (Smart), Penumbra Coil 400TM (PC 400), and Penumbra Occlusion Device (POD®). Data for each patient are collected in accordance with the standard of care at each participating hospital through one-year follow-up. Approximately 1,000 patients with intracranial aneurysms or other malformations treated by the Smart System at up to 100 centers will be enrolled. It is anticipated patient enrollment will take 3 years. All patients are to be assessed in accordance with the standard of care at each participating hospital through one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in this study must sign the Informed Consent Form and be treated according to the cleared indications for the Smart, PC 400, and POD, which include the embolization of:

* Intracranial aneurysms
* Other neurovascular abnormalities such as arteriovenous malformations and arteriovenous fistulae

Exclusion Criteria:

* Life expectancy less than one year
* Smart, PC 400, or POD account for less than 75% of total number of coils implanted
* Participation in another clinical investigation that could confound the evaluation of the registry device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 995 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (71):
  - Southeast Alabama Medical Center, Dothan, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - BNI, Phoenix, Arizona
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - Community Regional, Fresno, California
  - Loma Linda Medical Center, Loma Linda, California
  - Mercy San Juan, Sacramento, California
  - Cottage Hospital, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - RIA - Swedish Medical Center, Englewood, Colorado
  - St. Anthony's Hospital, Lakewood, Colorado
  - RIA - Lutheran Medical Center, Wheat Ridge, Colorado
  - Christiana Health, Newark, Delaware
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - CARE - Palmetto, Hialeah, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Jackson Memorial, Miami, Florida
  - Mt. Sinai Miami, Miami, Florida
  - Westside Regional Medical Center, Plantation, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - WellStar Kennestone Hospital, Marietta, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern Memorial, Chicago, Illinois
  - North Shore University, Evanston, Illinois
  - Clinical Radiologist, Springfield, Illinois
  - KUMC, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Metro Health Hospital, Wyoming, Michigan
  - HCMC, Minneapolis, Minnesota
  - UM-Fairview, Minneapolis, Minnesota
  - SSM Health Care, Fenton, Missouri
  - Overlook Medical Center, Summit, New Jersey
  - Kaleida Health, Buffalo, New York
  - UHS Wilson Medical Center, Johnson City, New York
  - Northshore, Manhasset, New York
  - Faxton St. Luke's Hospital, New Hartford, New York
  - Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - St. Vincent, Toledo, Ohio
  - OUHSC, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hershey's Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Palmetto Health, Columbia, South Carolina
  - Erlanger Health System, University of TN College of Medicine, Chattanooga, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist, Memphis, Tennessee
  - Baptist Hospital, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Houston Methodist, Houston, Texas
  - Texas Stroke Institute, Plano, Texas
  - Dept. of Neurosurgery, Univ of VA School of Medicine, Charlottesville, Virginia
  - Valley Health Winchester, Winchester, Virginia
  - Overlake Hospital, Bellevue, Washington
  - Tacoma General, Tacoma, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Royal University, Saskatoon, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashouri Y, Paul AR, AlMajali M, Chaudhari A, Lin E, Park MS, Bellon RJ, Bohnstedt BN, Yoo AJ, Schirmer CM, DeLeacy RA, Fiorella DJ, Woodward K, Hawk HE, Nanda A, Sunenshine PJ, Kabbani MR, Snyder KV, Sivapatham T, Dumont TM, Reeves AR, Starke RM, Spiotta AM, Zaidat OO. Large and giant intracranial aneurysms: outcomes from the multicenter prospective SMART coils registry. Front Neurol. 2026 Jan 14;16:1670622. doi: 10.3389/fneur.2025.1670622. eCollection 2025. PMID 41613189
- [Derived] Spiotta AM, Park MS, Bellon RJ, Bohnstedt BN, Yoo AJ, Schirmer CM, DeLeacy RA, Fiorella DJ, Woodward BK, Hawk HE, Nanda A, Zaidat OO, Sunenshine PJ, Liu KC, Kabbani MR, Snyder KV, Sivapatham T, Dumont TM, Reeves AR, Starke RM; SMART Registry Investigators. The SMART Registry: Long-Term Results on the Utility of the Penumbra SMART COIL System for Treatment of Intracranial Aneurysms and Other Malformations. Front Neurol. 2021 Apr 13;12:637551. doi: 10.3389/fneur.2021.637551. eCollection 2021. PMID 33927680
- [Derived] Starke RM, Park MS, Bellon R, Bohnstedt B, Schirmer CM, De Leacy R, Fiorella D, Yoo AJ, Spiotta AM; SMART Registry Investigators. Periprocedural safety of saccular aneurysm embolization with the Penumbra SMART Coil System: a SMART registry subset analysis. J Neurointerv Surg. 2022 Jan;14(1):neurintsurg-2020-016943. doi: 10.1136/neurintsurg-2020-016943. Epub 2021 Feb 16. PMID 33593799

RESULTS

PARTICIPANT FLOW:
Groups:
- Penumbra Smart System: Penumbra Smart Coil
  Penumbra Coil 400TM (PC400), Penumbra Occlusion DeviceTM(POD): Other Penumbra Coils available as standard of care
Period: Overall Study
Arm/Group | Penumbra Smart System
Started | 995
Completed | 864
Not Completed | 131
Not completed — Early Termination | 130
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Penumbra Smart System
Number analyzed (Participants) | 995
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 717
  Male | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall total because Ethnicity was captured later in the study.
  Participants
    number analyzed (Participants) | 326
    Hispanic or Latino | 33
    Not Hispanic or Latino | 293
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Number analyzed differs from overall total because Race was captured later in the study.
  Participants
    number analyzed (Participants) | 326
    American Indian or Alaska Native | 4
    Asian | 6
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 43
    White | 256
    More than one race | 0
    Unknown or Not Reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Adequate Occlusion Immediate Post Procedure
Description: Based on investigator's adjudication of adequate occlusion given anatomical and other considerations immediate post-procedure.
Time Frame: Immediate Post Procedure
Population: The analysis population (ITT) contains all 995 patients. 994 of 995 ITT patients have data on adequate occlusion at immediate post procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Smart System
Number analyzed (Participants) | 994
Participants | 965

2. Primary Outcome: Number of Times Re-access With Guidewire Was Required Due to Catheter Kickout
Description: Re-access attempts due to catheter kick-out across all coils
Time Frame: Immediate Post Procedure
Population: The analysis population is per device.
Measure: Number; unit: Coils
Units Other Than Participants: Coils
Arm/Group | Penumbra Smart System
Number analyzed (Participants) | 995
Number analyzed (Coils) | 5733
Coils | 317

3. Primary Outcome: Number of Procedural Device-related Serious Adverse Events at Immediate Post-procedure
Time Frame: Immediate Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Smart System
Number analyzed (Participants) | 995
Participants | 26

4. Primary Outcome: Number of Participants Requiring Retreatment Through Follow-up
Time Frame: One year from enrollment
Population: The number of participants analyzed is different from overall as these were subjects that returned for follow-up in the intent to treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Smart System
Number analyzed (Participants) | 784
Participants | 53

ADVERSE EVENTS:
Time Frame: 1 year
Description: Since this a post market registry, we will only be collecting Adverse Events (AEs) related to the procedure or device, unanticipated adverse device effects (UADE), and all Serious Adverse Events (SAEs) from the time of consent through registry exit. If an AE occurs that is not related to the procedure or device, it is not reportable under this Protocol.
Arm/Group | Penumbra Smart System
All-Cause Mortality (participants affected / at risk) | 60/995
Serious Adverse Events (participants affected / at risk) | 277/995
Other Adverse Events (participants affected / at risk) | 90/995
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra Smart System (N=995)
Anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 1
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial tachycardia (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 2
Cardiopulmonary failure (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Retinal hemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 7
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gastrointestinal ulcer (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Megacolon (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 3
Death (General disorders) | 5
Multiple organ dysfunction syndrome (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Vascular stent stenosis (General disorders) | 1
Vascular stent thrombosis (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Bacterial infection (Infections and infestations) | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haemophilus sepsis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 11
Sepsis (Infections and infestations) | 5
Septic shock (Infections and infestations) | 8
Staphylococcal infection (Infections and infestations) | 1
Thrombophlebitis septic (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Aneurysm recanalisation (Injury, poisoning and procedural complications) | 2
Brain herniation (Injury, poisoning and procedural complications) | 3
Face injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Incision site complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 13
Subdural haematoma (Injury, poisoning and procedural complications) | 5
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Vascular access site complication (Injury, poisoning and procedural complications) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Neurological examinations abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Lactic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Brain compression (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 8
Brain stem infarction (Nervous system disorders) | 1
Brain stem stroke (Nervous system disorders) | 1
Carotid artery aneurysm (Nervous system disorders) | 1
Carotid artery dissection (Nervous system disorders) | 5
Cerebral aneurysm perforation (Nervous system disorders) | 6
Cerebral artery embolism (Nervous system disorders) | 1
Cerebral artery occlusion (Nervous system disorders) | 5
Cerebral artery thrombosis (Nervous system disorders) | 3
Cerebral congestion (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 4
Cerebral infarction (Nervous system disorders) | 7
Cerebral thrombosis (Nervous system disorders) | 4
Cerebral vasoconstriction (Nervous system disorders) | 14
Cerebral venous thrombosis (Nervous system disorders) | 1
Cerebral ventricle dilatation (Nervous system disorders) | 1
Cerebral spinal fluid leakage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 1
Dural arteriovenous fistula (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 4
Haemorrhage intracranial (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 13
Hemiparesis (Nervous system disorders) | 3
Hydrocephalus (Nervous system disorders) | 23
Hypertensive encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 4
Intracranial pressure increased (Nervous system disorders) | 3
Ischaemic cerebral infarction (Nervous system disorders) | 3
Ischaemic stroke (Nervous system disorders) | 12
Migraine (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 3
Partial seizures (Nervous system disorders) | 1
Phantom pain (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 10
Seizure like phenomena (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 3
Subarachnoid hematoma (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 5
Transient global amnesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 7
VIth nerve paralysis (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Apathy (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Psychogenic seizure (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
End stage renal disease (Renal and urinary disorders) | 2
Renal injury (Renal and urinary disorders) | 1
Urethral haemorrhage (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary eodema (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cerebral endovascular aneurysm repair (Surgical and medical procedures) | 1
Peripheral artery stent insertion (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 6
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Intermittent claudication (Vascular disorders) | 1
Labile blood pressure (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 10
Venous stenosis (Vascular disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra Smart System (N=995)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 30
Nervous system disorders (Nervous system disorders) | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT02729740/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02729740/SAP_001.pdf